CLINICAL TRIAL: NCT07191704
Title: Characterization of Progressive Familial Intrahepatic Cholestasis (PFIC)-Related Genes in Adult Patients With Idiopathic Recurrent and Chronic Cholestasis in Spain - REGENIC
Brief Title: A Study to Assess the Genetic Variations in Bile Flow Disorders: Linking Progressive Familial Intrahepatic Cholestasis (PFIC)-Related Genes to Symptoms in Adults With Recurrent Cholestasis in Spain
Acronym: REGENIC
Status: Recruiting | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: CLIN-60240-453
Record Dates: First submitted 2025-09-17; First posted 2025-09-25 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: PFIC - Progressive Familial Intrahepatic Cholestasis
Keywords: Cholestasis
MeSH Terms: conditions — Cholestasis, progressive familial intrahepatic 1; Cholestasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Progressive Familial Intrahepatic Cholestasis (PFIC) is a group of inherited conditions that affect how bile moves in the liver, which can lead to serious liver problems. Doctors usually recommend genetic testing for patients with unexplained bile issues-after ruling out more common causes-to better understand the problem. However, there isn't much information on how common these genetic changes are in adults with these liver issues, especially in Spain. This study will observe these genetic changes so that doctors can diagnose the condition more clearly and create personalized treatment plans.

This study will be conducted in several centers across Spain for 10 months. Each adult participant will take part in a single-day visit where their health information will be collected, and a blood sample will be taken for both routine tests and genetic analysis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years old) with written informed consent prior to data collection and study procedures.
* Unexplained recurrent and/or chronic cholestasis (idiopathic cholestasis), defined as alkaline phosphatase (ALP) or Gamma-Glutamyl Transferase (GGT) > Upper Limit of Normal (ULN).
* Patients who provide the blood sample for the genetic analysis.

Exclusion Criteria:

* Patients with clear and confirmed diagnosed causes of cholestasis, including:

  * Primary Biliary Cholangitis
  * Primary or Secondary Sclerosing Cholangitis
  * Obstruction of the bile ducts
  * Other Liver diseases: cholestasis secondary to hepatocellular injury, viral hepatitis (mainly Hepatitis A virus [HAV], Hepatitis B virus [HBV] and Hepatitis C virus [HCV]), toxic hepatitis (pharmacological; drug-induced liver injury [DILI]), autoimmune hepatitis; intestinal failure, total parenteral nutrition [TPN]; Wilson's disease, choledochal cyst, Caroli Syndrome, and thick bile due to haemolysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 150 patients, both male and female, of age (≥ 18 years) with unexplained recurrent and/or chronic cholestasis (idiopathic cholestasis) will be recruited
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with at least One Variant in PFIC-Related Genes | At enrollment
  Defined as the percentage of participants with at least one variant in PFIC-related genes in relation to the total number of participants with idiopathic recurrent and/or chronic cholestasis of the study cohort as an assessment of prevalence.

SECONDARY OUTCOMES:
Percentage of Participants Carrying Each Identified Variant of Genes related to PFIC | At enrollment
  Defined as the percentage of participants carrying each identified variant of genes related to PFIC.
Demographic Data: Age at Enrollment | At enrollment
  Defined as the mean age of participants recorded at the time of enrollment, as noted in medical records, stratified by the PFIC type - comparing those with the most prevalent PFIC variant against all other participants.
Demographic Data: Sex at Enrollment | At enrollment
  Defined as the count of sex of participants recorded at the time of enrollment, as noted in medical records, stratified by the PFIC type - comparing those with the most prevalent PFIC variant against all other participants.
Demographic Data: Race/Ethnicity at Enrollment | At enrollment
  Defined as the race/ethnicity of participants recorded at the time of enrollment, as noted in medical records, stratified by the PFIC type - comparing those with the most prevalent PFIC variant against all other participants.
Demographic Data: Weight at Enrollment | At enrollment
  Defined as the mean weight participants recorded at the time of enrollment, as noted in medical records, stratified by the PFIC type - comparing those with the most prevalent PFIC variant against all other participants.
Demographic Data: Height at Enrollment | At enrollment
  Defined as the mean height participants recorded at the time of enrollment, as noted in medical records, stratified by the PFIC type - comparing those with the most prevalent PFIC variant against all other participants.
Demographic Data: Body Mass Index (BMI) at Enrollment | At enrollment
  Defined as the mean BMI, calculated by dividing participant's weight in kilograms by the square of their height in meters (BMI = weight ÷ height²), as noted in medical records, stratified by the PFIC type - comparing those with the most prevalent PFIC variant against all other participants.
Demographic Data: Alcohol Consumption at Enrollment | At enrollment
  Defined as the mean of standard drinks in a week to assess the alcohol consumption, recorded at the time of enrollment, as noted in medical records, stratified by the PFIC type - comparing those with the most prevalent PFIC variant against all other participants.
Age at Cholestasis Diagnosis | At enrollment
  Defined as the mean participant's age when first symptoms were reported, as noted in medical records or participant recollection, stratified by the PFIC type - comparing those with the most prevalent PFIC variant against all other participants.
History of Liver Disease | At enrollment
  Defined as the count of presence of liver conditions such as gallstones, pancreatitis, and cirrhosis (among other relevant conditions), as noted in medical records, stratified by the PFIC type - comparing those with the most prevalent PFIC variant against all other participants.
History of Diagnostic Procedures Used | At enrollment
  Defined as the count of presence of diagnostic procedures performed, including liver biopsy and elastography (Fibroscan) as noted in medical records, stratified by the PFIC type - comparing those with the most prevalent PFIC variant against all other participants.
Presence of Liver Disease Symptoms | At enrollment
  Defined as the count of presence of liver condition symptoms such as jaundice, pruritus and disease-related fatigue, as noted in medical records or participant recollection, stratified by the PFIC type - comparing those with the most prevalent PFIC variant against all other participants.
History of liver or biliary disease related surgeries | At enrollment
  Defined as the count of history of liver or biliary disease related surgeries, such as cholecystectomy, liver transplantation, surgical biliary diversion (SBD) or other liver-related surgery, as noted in medical records, stratified by the PFIC type - comparing those with the most prevalent PFIC variant against all other participants.
Family history of liver disease | At enrollment
  Defined as the count of family history of liver disease, such as the presence or absence of PFIC, intrahepatic cholestasis of pregnancy (ICP), benign recurrent intrahepatic cholestasis (BRIC), low-phospholipid-associated cholelithiasis (LPAC), portal hypertension, hepatocellular carcinoma, cholangiocarcinoma, pancreatitis, gallstones, cirrhosis, cholestatic drug induced liver injury (DILI), Metabolic dysfunction-associated fatty liver disease (MASLD), Non-alcoholic Steatohepatitis (MASH) and any other chronic liver disease, and which close relative has suffered it (parent, grandparent, sibling, etc.), as noted in medical records or participant recollection, stratified by the PFIC type - comparing those with the most prevalent PFIC variant against all other participants.
Presence or Absence of Fat-Soluble Vitamin deficiencies | At enrollment
  Defined as the count of presence or absence of vitamin deficiencies, such as vitamin A, D, E and K and supplementation, as noted in medical records or participant recollection, stratified by the PFIC type - comparing those with the most prevalent PFIC variant against all other participants.
Laboratory Analysis of Haematology - Haemoglobin | At enrollment
  Defined as the last recorded routine analysis of haemoglobin, stratified by the PFIC type - comparing those with the most prevalent PFIC variant against all other participants.
Laboratory Analysis of Haematology - Red Blood Cell (RBC) count | At enrollment
  Defined as the last recorded routine analysis of RBC count, as noted in medical records, stratified by the PFIC type - comparing those with the most prevalent PFIC variant against all other participants.
Laboratory Analysis of Haematology - Leukocytes | At enrollment
  Defined as the last recorded routine analysis of leukocytes, as noted in medical records, stratified by the PFIC type - comparing those with the most prevalent PFIC variant against all other participants.
Laboratory Analysis of Haematology - Platelets | At enrollment
  Defined as the last recorded routine analysis of platelets, as noted in medical records, stratified by the PFIC type - comparing those with the most prevalent PFIC variant against all other participants.
Laboratory Analysis of Chemistry - Alanine aminotransferase (ALT) | At enrollment
  Defined as the recorded routine analysis of ALT, as noted in medical records, stratified by the PFIC type - comparing those with the most prevalent PFIC variant against all other participants.
Laboratory Analysis of Chemistry - Aspartate aminotransferase (AST) | At enrollment
  Defined as the recorded routine analysis of AST, as noted in medical records, stratified by the PFIC type - comparing those with the most prevalent PFIC variant against all other participants.
Laboratory Analysis of Chemistry - Alkaline Phosphatase (ALP) | At enrollment
  Defined as the recorded routine analysis of ALP, as noted in medical records, stratified by the PFIC type - comparing those with the most prevalent PFIC variant against all other participants.
Laboratory Analysis of Chemistry - Total and direct bilirubin | At enrollment
  Defined as the recorded routine analysis of total and direct bilirubin, as noted in medical records, stratified by the PFIC type - comparing those with the most prevalent PFIC variant against all other participants.
Laboratory Analysis of Chemistry - Bile Acids (sBA) | At enrollment
  Defined as the recorded routine analysis of sBA, as noted in medical records, stratified by the PFIC type - comparing those with the most prevalent PFIC variant against all other participants.
Laboratory Analysis of Chemistry - Gamma-Glutamyl Transferase (GGT) | At enrollment
  Defined as the recorded routine analysis of GGT, as noted in medical records, stratified by the PFIC type - comparing those with the most prevalent PFIC variant against all other participants.
Laboratory Analysis of Chemistry - Albumin | At enrollment
  Defined as the recorded routine analysis of albumin, as noted in medical records, stratified by the PFIC type - comparing those with the most prevalent PFIC variant against all other participants.
Laboratory Analysis of Coagulation - Prothrombin time | At enrollment
  Defined as the recorded routine analysis of prothrombin time, as noted in medical records, stratified by the PFIC type - comparing those with the most prevalent PFIC variant against all other participants.
Laboratory Analysis of Coagulation - International Normalized Ratio (INR) | At enrollment
  Defined as the recorded routine analysis of INR, as noted in medical records, stratified by the PFIC type - comparing those with the most prevalent PFIC variant against all other participants.
Frequency of Prior and Concomitant treatment for cholestatic liver disease and pruritus. | At enrollment
  Defined as the count of prior and concomitant treatment for cholestatic liver disease and pruritus: ursodeoxycholic acid (UDCA), cholestyramine, rifampicin, fibrates, ileal bile acid transporter inhibitors (IBATi), selective serotonin reuptake inhibitors (SSRI), opioid antagonists, Chaperones (4- phenylbutyrate, [4-PB]) skin emollients or others, as noted in medical records or participant recollection, stratified by the PFIC type - comparing those with the most prevalent PFIC variant against all other participants.
Comorbidities of interest (i.e., diabetes, metabolic syndrome, osteopenia/osteoporosis) | At enrollment
  Defined as the count of comorbidities of interest, such as diabetes, metabolic syndrome, osteopenia/osteoporosis, as noted in medical records or participant recollection, stratified by the PFIC type - comparing those with the most prevalent PFIC variant against all other participants.

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (10):
- Spain (10):
  - H. Clinic (first CEIm), Barcelona
  - H. Vall Hebron, Barcelona
  - H. Reina Sofía, Córdoba
  - H. Dr. Negrín, Las Palmas
  - H. Gregorio Marañón, Madrid
  - Hospital Universitario La Paz, Madrid
  - H. Virgen del Rocío, Seville
  - H. La Fe, Valencia
  - H. Río Hortega, Valladolid
  - H. Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications.
  Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and/or EU.
Access Criteria: Further details on Ipsen's sharing criteria and process for sharing are available here (https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/).
URL: https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/